CLINICAL TRIAL: NCT02816489
Title: A Randomized Clinical Trial to Evaluate Labial Alveolar Bone Thickness and Apical Root Resorption Between Two Kinds of Brackets Using CBCT
Brief Title: Labial Alveolar Bone Thickness and Apical Root Resorption Changes Associated With Self-ligating Versus Conventional Brackets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 9046380
Record Dates: First submitted 2016-05-30; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Labial Alveolar Bone Thickness; Apical Root Resorption

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): will be treated using passive self-ligating ceramic orthodontic brackets with stainless steel archwire slot liner (3M Unitek - USA).
  Intervention: Device: passive self-ligating ceramic orthodontic brackets with stainless steel archwire slot liner (3M Unitek - USA).
  Interventions: Device: Clarity SL MBT brackets; 3M Unitek, Monrovia, CA, USA
- Group II (Experimental): will be treated using conventional stainless steel orthodontic brackets ligated with elastomeric ligature (3M Unitek - USA).
  Intervention: Device: conventional stainless steel orthodontic brackets ligated with elastomeric ligature (3M Unitek - USA).
  Interventions: Device: Gemini MBT brackets; 3M Unitek, Monrovia, CA, USA

INTERVENTIONS:
Device: Clarity SL MBT brackets; 3M Unitek, Monrovia, CA, USA — (passive self-ligating ceramic orthodontic brackets with stainless steel archwire slot liner)
  Other Names: Clarity SL
  Arms: Group I
Device: Gemini MBT brackets; 3M Unitek, Monrovia, CA, USA — (conventional stainless steel orthodontic brackets ligated with elastomeric ligature)
  Other Names: Gemini
  Arms: Group II

SUMMARY:
Labial alveolar bone thickness and apical root resorption changes associated with self-ligating versus conventional brackets.

The aim of this study will be to compare labial alveolar bone thickness and apical root resorption changes associated with self-ligating versus conventional brackets.

DETAILED DESCRIPTION:
Labial alveolar bone thickness and apical root resorption changes associated with self-ligating versus conventional brackets.

Protocol submitted in partial fulfillment for the requirements of Master Degree in Orthodontics.

The initial stage of treatment crowding permanent teeth orthodontically is worried about teeth leveling and alignment. The accuracy of this procedure depends on various variables.

Friction is generated upon the materialistic composition of different bracket and archwire types, and the technique of ligature between them.

Several self-ligating brackets have been grown since 1935. Self-ligation doesn't need for an elastomeric attachment to catch the archwire, so it is related with a highly reduced friction with many different types of archwires, therefore less force required.

It is valuable to evaluate any appliance system for its capability to align teeth with minimal injurious effects to the oral tissues.

The aim of this study will be to compare labial alveolar bone thickness and apical root resorption changes associated with self-ligating versus conventional brackets.

Subjects and method

Study design:

Randomized controlled clinical trial

Study setting and population:

The sample of this study will be consisted of twenty one patients selected from Outpatient Clinic, Orthodontic Department, Faculty of Dentistry, Mansoura University.

Interventions:

The patients will be divided randomly into two groups and will be treated separately as follows:

* Group I: will be treated using passive self-ligating ceramic orthodontic brackets with stainless steel archwire slot liner.
* Group II: will be treated using conventional stainless steel orthodontic brackets ligated with elastomeric ligature.

The patients will be treated orthodontically within the initial leveling and alignment for the 6 month duration beginning with the same sequence of 0.014, 0.016, 0.016 × 0.022 inch nickel-titanium archwires and 0.016 × 0.022 inch stainless-steel archwire. Each archwire will be remained for 1.5 months, and it will be replaced with the previously mentioned sequence. For group II, the archwires will be attached to the brackets by using an elastomeric ligature. CBCT will be obtained in two time intervals, before beginning the orthodontic treatment and 6 months after it. Dental stripping and extraction of premolars will be eliminated.

Records:

For all patients the following records will be taken before and after leveling and alignment:

1. Standardized upper and lower study casts.
2. Standardized periapical radiograph.
3. Standardized extra-oral and intra-oral photographs.
4. Standardized cone beam computed tomography (CBCT).

Observations:

Sagittal cuts of upper and lower incisors in the center of the long axis will be selected. The labial alveolar bone thickness (LABT) of each incisor will be determined at the site neighboring to the widest point of the labiopalatal root in two levels separated by 3 mm (L1 and L2, respectively); these levels will be set along the long axis of the incisor and located every 3 mm from the cementoenamel junction (CEJ) level. Labial alveolar bone thickness will be assessed at the cervical level (L1) and midroot level (L2) at T0 and T1. Furthermore, the apical root resorption (ARR) will be calculated by determining the difference in the total tooth length, which will be measured in millimeters from the incisal border to the root apex, between T0 and T1 (T1-T0).

Ethical consideration:

All patients will receive information about the future clinical trial study and give their consent by signing an informed consent.

Data management and analysis: All statistical analysis will be performed with SPSS software. Differences will be considered significant at P values less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranged between 14-20 years.
2. Complete permanent dentition (excluding third molars).
3. Angle Class I malocclusion.
4. Crowding anteriorly ranging from 2 to 4 mm.
5. Healthy young patients.

Exclusion Criteria:

1. Patients with signs of apical root resorption detected at the first examination by periapical radiographs.
2. Blocked-out or High-up canines.
3. Patients who went to previous orthodontic treatment.
4. Evidence of periodontal or gingival problems.
5. Endodontic treatment.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Labial alveolar bone thickness | Change from baseline in Labial alveolar bone thickness at 6 months
  Labial alveolar bone thickness will be measured in millimeters using CBCT at the site neighboring to the widest point of the labiopalatal root in two levels separated by 3 mm (L1 and L2, respectively); these levels were set along the long axis of the incisor and located every 3 mm from the cementoenamel junction (CEJ) level. Labial alveolar bone thickness was assessed at the cervical level (L1) and midroot level (L2) at T0 and T1.
Apical root resorption | Change from baseline in Apical root resorption at 6 months
  Apical root resorption will be measured in millimeters using CBCT by determining the difference in the total tooth length, which was measured from the incisal border to the root apex, between T0 and T1 (T1-T0).

CONTACTS AND LOCATIONS:
Locations (1):
- Al Mansurah, Egypt